CLINICAL TRIAL: NCT03386578
Title: Pharmacokinetics, Feasibility, Acceptability, and Safety of Oral Pre-Exposure Prophylaxis for Primary HIV Prevention During Pregnancy and Postpartum in Adolescents and Young Women and Their Infants
Brief Title: Evaluating the Pharmacokinetics, Feasibility, Acceptability, and Safety of Oral Pre-Exposure Prophylaxis for HIV Prevention During Pregnancy and Postpartum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMPAACT 2009; 30020 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-12-18; First posted 2017-12-29 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Maternal PK Component Group 1 (Experimental): Mothers enrolled during singleton pregnancy at 14-24 weeks' gestation received PrEP once daily under direct observation from day 0 through week 12.
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF)
- Maternal PK Component Group 2 (Experimental): Mothers enrolled postpartum within 6-12 weeks after delivery received PrEP once daily under direct observation from day 0 through week 12.
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF)
- Maternal PrEP Comparison Cohort 1 (Experimental): Mothers who initiated PrEP at study entry received daily oral PrEP, a behavioral HIV risk reduction package and enhanced adherence support from day 0 through postpartum week 26.
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF); Behavioral: Behavioral HIV risk reduction package; Behavioral: Enhanced adherence support
- Maternal PrEP Comparison Cohort 2/Step 1 (Active Comparator): Mothers who declined PrEP initiation at study entry received a behavioral HIV risk reduction package from day 0 through postpartum week 26.
  Interventions: Behavioral: Behavioral HIV risk reduction package
- Maternal PrEP Comparison Cohort 2/Step 2 (Experimental): Mothers from Cohort 2/Step 1 who subsequently chose to initiate PrEP during the study received daily oral PrEP and enhanced adherence support from Step 2 entry through postpartum week 26, along with the behavioral HIV risk reduction package.
  Interventions: Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF); Behavioral: Behavioral HIV risk reduction package; Behavioral: Enhanced adherence support
- Infant PK Component Group 1 (No Intervention): Infants born to women in PK Component Group 1. Infants did not directly receive PrEP, but may have been exposed to PrEP through placental or breastmilk transfer.
- Infant PK Component Group 2 (No Intervention): Infants born to women in PK Component Group 2. Infants did not directly receive PrEP, but may have been exposed to PrEP through breastmilk transfer.
- Infant PrEP Comparison Cohort 1 (No Intervention): Infants born to women in PrEP Comparison Cohort 1. Infants did not directly receive PrEP, but may have been exposed to PrEP through placental or breastmilk transfer.
- Infant PrEP Comparison Cohort 2/Step 1 (No Intervention): Infants born to women in PrEP Comparison Cohort 2/Step 1. Infants were not exposed to PrEP during the study.
- Infant PrEP Comparison Cohort 2/Step 2 (No Intervention): Infants born to women in PrEP Comparison Cohort 2/Step 2. Infants did not directly receive PrEP, but may have been exposed to PrEP through placental or breastmilk transfer.

INTERVENTIONS:
Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) — 200 mg/300 mg of FTC/TDF administered orally as a fixed-dose combination tablet once daily
  Other Names: Truvada
  Arms: Maternal PK Component Group 1; Maternal PK Component Group 2; Maternal PrEP Comparison Cohort 1; Maternal PrEP Comparison Cohort 2/Step 2
Behavioral: Behavioral HIV risk reduction package — Included cohort-appropriate SMS messages.
  Arms: Maternal PrEP Comparison Cohort 1; Maternal PrEP Comparison Cohort 2/Step 1; Maternal PrEP Comparison Cohort 2/Step 2
Behavioral: Enhanced adherence support — Included two-way SMS messaging and tailored counseling with drug level feedback.
  Arms: Maternal PrEP Comparison Cohort 1; Maternal PrEP Comparison Cohort 2/Step 2

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetics, feasibility, acceptability, and safety of a fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate (FTC/TDF) as oral daily pre-exposure prophylaxis (PrEP) to prevent HIV during pregnancy and postpartum in adolescents and young women and their infants.

DETAILED DESCRIPTION:
This study evaluated the pharmacokinetics, feasibility, acceptability, and safety of FTC/TDF as oral daily PrEP to prevent HIV during pregnancy and postpartum in adolescents and young women and their infants. The study was conducted in two consecutive components: 1) Pharmacokinetics (PK) Component and 2) PrEP Comparison Component.

In the PK Component, women enrolled in one of two groups. Group 1 included pregnant women at 14 to 24 weeks' gestation and Group 2 included postpartum women who delivered 6 to 12 weeks prior to enrollment. Both groups received a fixed-dose combination of FTC/TDF administered once daily by direct observation from Day 0 through Week 12.

Mothers in the PK Component had weekly study visits through Week 12. Infants in Group 1, whose mothers enrolled during pregnancy, had study visits at birth and six weeks of life; infants in Group 2, who were enrolled with their mothers 6-12 weeks after birth, had study visits at Week 6 and Week 12. Study visits for mothers and infants in the PK Component included evaluation of drug levels and monitoring for adverse effects.

In the PrEP Comparison Component, pregnant women enrolled in one of two cohorts. Mothers in Cohort 1 chose to initiate PrEP at study entry, and mothers in Cohort 2 declined PrEP at entry. Participants in both Cohorts received a standard of care package of HIV prevention services, a study-specific behavioral risk reduction intervention, and periodic one-way short message service (SMS) messages to promote maternal and child health from Day 0 through Week 26. Cohort 1 opted to also receive daily oral FTC/TDF as PrEP and enhanced adherence support, including weekly two-way SMS messaging and feedback of drug levels with tailored adherence counseling. Participants who changed their mind about using PrEP during study participation were able to subsequently stop PrEP (Cohort 1) or initiate PrEP (Cohort 2/Step 2).

Mothers in the PrEP Comparison Component had regular study visits through delivery and Week 26 (postpartum). Infants in the PrEP Comparison Component had four study visits from birth through week 26 of life. For mothers, study visits included physical examinations, blood and urine collection, vaginal and (optional) rectal swab collection, vaginal secretions collection, ultrasounds, and dual-energy x-ray absorptiometry (DXA) scans. For infants, study visits included physical examinations, rectal swab and blood collection, and DXA scans.

In the PrEP Comparison Component analysis, maternal and infant participants were classified based on their PrEP exposure. The PrEP-exposed group included participants from Cohort 1 (throughout the entire study follow-up) and from Cohort 2/Step 2 (from Step 2 entry to the end of follow-up). The PrEP-unexposed group comprised participants from Cohort 2/Step 1 who did not enroll in Cohort 2/Step 2 (throughout the entire study follow-up) or who enrolled in Cohort 2/Step 2 (from study entry until enrolling in Cohort 2/Step 2).

ELIGIBILITY:
PK Component (Groups 1 and 2) Inclusion Criteria:

* At study entry, pregnant or recently delivered, in one of the following two enrollment windows:

  * Group 1: Gestational age of 14 to 24 weeks.
  * Group 2: 6 to 12 weeks postpartum.
* Willing to initiate daily PrEP for 12 weeks under directly observed therapy.
* HIV and Hepatitis B negative.
* At screening:

  * Grade 1 or normal alanine transaminase (ALT), hemoglobin (HB), absolute neutrophil count (ANC) and normal creatinine clearance (CrCl).
  * Negative or trace proteinuria (less than Grade 1).
  * Normal dipstick urine for glucose (less than Grade 1).
  * Mother weighs greater than 35 kg.
* Intention to stay within the study site's catchment area for at least 12 weeks (or through delivery).

Exclusion Criteria (PK Component and PrEP Comparison Component):

* Any current significant uncontrolled, active or chronic disease process.
* History of any of the following:

  * Sickle cell anemia, chronic bleeding, blood transfusion within the past 120 days or other blood dyscrasias
  * Bone fracture not explained by trauma
  * Allergy/sensitivity to FTC/TDF or its components
* Fetus has a known or suspected major congenital anomaly
* Mother has confirmed renal insufficiency, a history of renal parenchymal disease or single kidney
* Current use of prohibited medications listed in the protocol
* Concurrent participation in any biomedical HIV prevention or investigational drug in an HIV vaccine or microbicide study
* Past participation in an HIV vaccine study
* Currently taking a PrEP regimen from non-study sources
* Any other condition or adverse social situation
* Past participation in IMPAACT 2009

PrEP Comparison Component (Cohorts 1 and 2) Inclusion Criteria:

* At screening, evidence of a viable singleton pregnancy with gestational age of 32 weeks or less.
* Within 14 days prior to study entry, negative HIV RNA test.
* HIV and Hepatitis B negative.
* At screening:

  * Grade 1 or normal ALT, HB, ANC and normal CrCl.
  * Negative or trace proteinuria (less than Grade 1).
  * Normal dipstick urine for glucose (less than Grade 1).
* Intention to stay within the study site's catchment area through 26 weeks postpartum
* A cellular phone that is able to receive SMS messages, and for Cohort 1 only, is also able to send SMS messages.
* Cohort 1 only: Willingness to take PrEP from pregnancy up to 26 weeks postpartum
* Cohort 2 only: Unwillingness to take PrEP from pregnancy up to 26 weeks postpartum
* Mother weighs greater than 35 kg
* Mother is literate in one or more of the study languages

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 780 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2024-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chi, MD, MSc, Study Chair — University of North Carolina, Chapel Hill; Lynda Stranix-Chibanda, MBChB, MMED, Study Chair — University of Zimbabwe Faculty of Medicine and Health Sciences
Locations (7):
- Blantyre CRS, Blantyre, Malawi
- Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng, South Africa
- Uganda (2):
  - Baylor-Uganda CRS, Kampala
  - MU-JHU Care Limited CRS, Kampala
- Zimbabwe (3):
  - St Mary's CRS, Saint Mary's, Chitungwiza
  - Seke North CRS, Chitungwiza
  - Harare Family Care CRS, Harare

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.

REFERENCES:
- [Result] Stranix-Chibanda L, Anderson PL, Kacanek D, Hosek S, Huang S, Nematadzira TG, Taulo F, Korutaro V, Nakabiito C, Masenya M, Lypen K, Brown E, Ibrahim ME, Yager J, Wiesner L, Johnston B, Amico KR, Rooney JF, Chakhtoura N, Spiegel HML, Chi BH; IMPAACT 2009 Team. Tenofovir Diphosphate Concentrations in Dried Blood Spots From Pregnant and Postpartum Adolescent and Young Women Receiving Daily Observed Pre-exposure Prophylaxis in Sub-Saharan Africa. Clin Infect Dis. 2021 Oct 5;73(7):e1893-e1900. doi: 10.1093/cid/ciaa1872. PMID 33341883
- See also: Related Info — http://impaactnetwork.org/studies/IMPAACT2009.asp
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Period: PK Component
Arm/Group | Maternal PK Component Group 1 | Maternal PK Component Group 2 | Maternal PrEP Comparison Cohort 1 | Maternal PrEP Comparison Cohort 2/Step 1 | Maternal PrEP Comparison Cohort 2/Step 2 | Infant PK Component Group 1 | Infant PK Component Group 2 | Infant PrEP Comparison Cohort 1 | Infant PrEP Comparison Cohort 2/Step 1 | Infant PrEP Comparison Cohort 2/Step 2
Started | 20 | 20 | 0 | 0 | 0 | 20 | 20 | 0 | 0 | 0
Completed | 20 | 19 | 0 | 0 | 0 | 18 | 19 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Stillbirth/Abortion | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: PrEP Comparison Component Step 1
Arm/Group | Maternal PK Component Group 1 | Maternal PK Component Group 2 | Maternal PrEP Comparison Cohort 1 | Maternal PrEP Comparison Cohort 2/Step 1 | Maternal PrEP Comparison Cohort 2/Step 2 | Infant PK Component Group 1 | Infant PK Component Group 2 | Infant PrEP Comparison Cohort 1 | Infant PrEP Comparison Cohort 2/Step 1 | Infant PrEP Comparison Cohort 2/Step 2
Started | 0 | 0 | 229 | 121 | 0 | 0 | 0 | 229 | 121 | 0
Completed | 0 | 0 | 202 | 95 | 0 | 0 | 0 | 196 | 88 | 0
Not Completed | 0 | 0 | 27 | 26 | 0 | 0 | 0 | 33 | 33 | 0
Not completed — Lost to Follow-up | 0 | 0 | 17 | 9 | 0 | 0 | 0 | 7 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 9 | 4 | 0 | 0 | 0 | 5 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 9 | 5 | 0
Not completed — Enrolled to Cohort 2/Step 2 | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0 | 13 | 0
Not completed — Stillbirth/Abortion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0
Not completed — Maternal Off-study During Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 5 | 0
Period: PrEP Comparison Component Step 2
Arm/Group | Maternal PK Component Group 1 | Maternal PK Component Group 2 | Maternal PrEP Comparison Cohort 1 | Maternal PrEP Comparison Cohort 2/Step 1 | Maternal PrEP Comparison Cohort 2/Step 2 | Infant PK Component Group 1 | Infant PK Component Group 2 | Infant PrEP Comparison Cohort 1 | Infant PrEP Comparison Cohort 2/Step 1 | Infant PrEP Comparison Cohort 2/Step 2
Started | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0 | 13
Completed | 0 | 0 | 0 | 0 | 13 | 0 | 0 | 0 | 0 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In the PrEP Comparison Component, baseline characteristics are summarized at enrollment into Cohort 1 or Cohort 2/Step 1. The study was primarily designed to enroll pregnant women, with infants being born during the course of the study. Therefore, the baseline analysis population only includes pregnant women at the time of enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maternal PK Component Group 1 | Maternal PK Component Group 2 | Maternal PrEP Comparison Cohort 1 | Maternal PrEP Comparison Cohort 2/Step 1 | Maternal PrEP Comparison Cohort 2/Step 2 | Total
Number analyzed (Participants) | 20 | 20 | 229 | 121 | 0 | 390
Age, Continuous [Median (Full Range); unit: years] — Population: Baseline age is reported separately for PK Component and PrEP Comparison Component participants.
  years
    PK Component: number analyzed (Participants) | 20 | 20 | 0 | 0 | 0 | 40
    PK Component | 20 [16 to 24] | 20 [16 to 23] |  |  |  | 20 [16 to 24]
    PrEP Comparison: number analyzed (Participants) | 0 | 0 | 229 | 121 | 0 | 350
    PrEP Comparison |  |  | 21 [17 to 24] | 21 [16 to 24] |  | 21 [16 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 229 | 121 | 0 | 390
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 20 | 20 | 229 | 121 | 0 | 390
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 0 | 7 | 23 | 27 |  | 57
  South Africa | 4 | 0 | 29 | 11 |  | 44
  Uganda | 8 | 4 | 54 | 23 |  | 89
  Zimbabwe | 8 | 9 | 123 | 60 |  | 200
Gestational Age [Median (Full Range); unit: weeks] — Population: Baseline gestational age is reported separately for PK Component and PrEP Comparison Component participants. PK Component Group 2 participants were enrolled during postpartum.
  weeks
    PK Component: number analyzed (Participants) | 20 | 0 | 0 | 0 | 0 | 20
    PK Component | 18 [11 to 23] |  |  |  |  | 18 [11 to 23]
    PrEP Comparison: number analyzed (Participants) | 0 | 0 | 229 | 121 | 0 | 350
    PrEP Comparison |  |  | 24 [9 to 31] | 25 [12 to 31] |  | 24 [9 to 31]

OUTCOME MEASURES:

1. Primary Outcome: Estimated Threshold of Maternal Steady-state Tenofovir Diphosphate (TFV-DP) Concentration Levels Corresponding to Optimal Adherence in the PK Component
Description: TFV-DP concentration levels were measured using dried blood spots (DBS) collected weekly during pregnancy and postpartum. These concentrations accumulated each week, and the plateau observed in the concentration-time curve represents the steady-state TFV-DP concentration, achieved at week 12. Predicted TFV-DP concentration levels for each maternal participant were obtained using a population PK model, and descriptive statistics were generated. The estimated steady-state TFV-DP concentration threshold for optimal adherence during pregnancy and postpartum is the 25th percentile when taking 7 doses per week. For more details, refer to the published paper (PubMed ID: 33341883).
Time Frame: Measured from study week 1 to study week 12 during pregnancy for Maternal PK Component Group 1 and from study week 1 to study week 12 during postpartum for Maternal PK Component Group 2
Population: Mothers from PK Component were included in this outcome measure.
Measure: Number; unit: fmol/punch
Arm/Group | Maternal PK Component Group 1 | Maternal PK Component Group 2
Number analyzed (Participants) | 20 | 20
fmol/punch | 965 | 1050

2. Primary Outcome: Proportion of Mothers With Optimal Adherence at Antepartum Study Week 4
Description: TFV-DP concentration levels were measured using dried blood spots (DBS). Mothers with optimal adherence were identified based on TFV-DP concentration levels and the threshold established in the PK Component.
Time Frame: Antepartum study week 4
Population: Mothers from the PrEP Comparison PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) who were formally prescribed PrEP and had available PK data were included in this analysis. All primary analyses, as described in the SAP, were conducted by two groups: PrEP-exposed and PrEP-unexposed. Cohort 1 and Cohort 2/Step 2 together were defined as the PrEP-exposed group and were analyzed together.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2): Cohort 1: Mothers who initiated PrEP at study entry received daily oral PrEP, a behavioral HIV risk reduction package and enhanced adherence support from day 0 through postpartum week 26.
  Cohort 2/Step 2: Mothers from Cohort 2/Step 1 who subsequently chose to initiate PrEP during the study received daily oral PrEP and enhanced adherence support from Step 2 entry through postpartum week 26, along with the behavioral HIV risk reduction package.
- Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1): Cohort 2/Step 1: Mothers who declined PrEP initiation at study entry received a behavioral HIV risk reduction package from day 0 through postpartum week 26.
Arm/Group | Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 194 | 0
proportion of participants | 0.15 [0.11 to 0.21] |

3. Primary Outcome: Proportion of Mothers With Optimal Adherence at Antepartum Study Week 8
Description: as for outcome 2
Time Frame: Antepartum study week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- PrEP Comparison: PrEP Exposed (Cohort 1 and Cohort 2/Step 2): Cohort 1: Mothers who initiated PrEP at study entry received daily oral PrEP, a behavioral HIV risk reduction package and enhanced adherence support from day 0 through postpartum week 26.
  Cohort 2/Step 2: Mothers from Cohort 2/Step 1 who subsequently chose to initiate PrEP during the study received daily oral PrEP and enhanced adherence support from Step 2 entry through postpartum week 26, along with the behavioral HIV risk reduction package.
- PrEP Comparison: PrEP Unexposed (Cohort 2/Step 1): Cohort 2/Step 1: Mothers who declined PrEP initiation at study entry received a behavioral HIV risk reduction package from day 0 through postpartum week 26.
Arm/Group | PrEP Comparison: PrEP Exposed (Cohort 1 and Cohort 2/Step 2) | PrEP Comparison: PrEP Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 159 | 0
proportion of participants | 0.23 [0.16 to 0.30] |

4. Primary Outcome: Proportion of Mothers With Optimal Adherence at Antepartum Study Week 12
Description: as for outcome 2
Time Frame: Antepartum study week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 95 | 0
proportion of participants | 0.27 [0.19 to 0.37] |

5. Primary Outcome: Proportion of Mothers With Optimal Adherence at Delivery
Description: as for outcome 2
Time Frame: Delivery
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 143 | 0
proportion of participants | 0.31 [0.23 to 0.39] |

6. Primary Outcome: Proportion of Mothers With Optimal Adherence at Postpartum Week 6
Description: as for outcome 2
Time Frame: Postpartum Week 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 168 | 0
proportion of participants | 0.20 [0.14 to 0.27] |

7. Primary Outcome: Proportion of Mothers With Optimal Adherence at Postpartum Week 14
Description: as for outcome 2
Time Frame: Postpartum week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 161 | 0
proportion of participants | 0.17 [0.12 to 0.24] |

8. Primary Outcome: Proportion of Mothers With Optimal Adherence at Postpartum Week 26
Description: as for outcome 2
Time Frame: Postpartum Week 26
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 110 | 0
proportion of participants | 0.15 [0.09 to 0.23] |

9. Primary Outcome: Proportion of Maternal Visits With Optimal Adherence During Study Follow-up
Description: as for outcome 2
Time Frame: Study entry through 26 weeks postpartum, up to one year
Population: Mothers from the PrEP Comparison PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) with PK data from any study visits were included in this analysis. All primary analyses, as described in the SAP, were conducted by two groups: PrEP-exposed and PrEP-unexposed. Cohort 1 and Cohort 2/Step 2 together were defined as the PrEP-exposed group and were analyzed together.
Measure: Number (95% Confidence Interval); unit: proportion of visits
Units Other Than Participants: Visits
Arm/Group | Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 219 | 0
Number analyzed (Visits) | 1032 | 0
proportion of visits | 0.21 [0.18 to 0.23] |

10. Primary Outcome: Incidence Rate of Maternal Adverse Events Per 100 Person-years
Description: Adverse events (AEs) were graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. Maternal AEs were defined as the occurrence of at least one grade 2 (moderate) chemistry abnormality, or one grade 3 (severe), grade 4 (potentially life-threatening), or grade 5 (death) adverse event, during the study follow-up.
Time Frame: Study entry through 26 weeks postpartum, up to one year
Population: Mothers from the PrEP Comparison Component were included in the analysis. Primary analyses, as described in the SAP, were conducted in two groups: PrEP-exposed and PrEP-unexposed. Cohort 1 and Cohort 2/Step 2 were combined as the PrEP-exposed group. The incidence of adverse events was calculated per 100 person-years. Maternal participants in Cohort 2/Step 2 contributed to person-years for both groups, with Cohort 2/Step 1 censored upon enrollment in Step 2.
Measure: Number (95% Confidence Interval); unit: number of new cases per 100 person years
Arm/Group | Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 242 | 121
number of new cases per 100 person years | 29.4 [22.1 to 36.0] | 18.2 [11.0 to 30.2]
Statistical Analysis 1: Comparison: Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); The incidence rate ratio of cumulative maternal adverse events was calculated between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and the PrEP-unexposed (Cohort 2/Step 1) reference group based on incidence per person-time follow-up. Maternal participants in Cohort 2/Step 2 contributed person-time to both Cohort 2/Step 1 and Step 2; Test type: Other; Incidence rate ratio = 1.62, 95% CI 2-sided [0.89 to 2.94]

11. Primary Outcome: Number of Composite Adverse Pregnancy Outcomes
Description: Adverse outcomes are defined as at least one of the following: spontaneous abortion (less than 20 weeks gestation), stillbirth (greater than or equal to 20 weeks gestation), preterm delivery (less than 37 weeks), or small for gestational age (less than 10th percentile using INTERGROWTH-21 norms)
Time Frame: Measured at delivery
Population: Mothers from PrEP Comparison Component with available pregnancy outcome data were included in this analysis. All primary analyses, as described in the SAP, were conducted by two groups: PrEP-exposed and PrEP-unexposed. Cohort 1 and Cohort 2/Step 2 together were defined as the PrEP-exposed group and were analyzed together.
Measure: Number; unit: participants
Arm/Group | Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 216 | 108
participants | 51 | 28
Statistical Analysis 1: Comparison: Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); Odds ratio comparing the proportion of mothers with adverse pregnancy outcomes between the PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed (Cohort 2/Step 1) reference group; Test type: Other; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.52 to 1.50]
Statistical Analysis 2: Comparison: Maternal PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Maternal PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); Test the differences in the proportion of mothers with adverse pregnancy outcomes between PrEP-exposed (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed (Cohort 2/Step 2) groups; Test type: Other; p = 0.68, Fisher Exact

12. Primary Outcome: Incidence Rate of Infant Grade 3 or Higher Adverse Events Per 100 Person-years
Description: Adverse events were assessed according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. An infant grade 3 or higher adverse event was defined as a grade 3 (severe), grade 4 (potentially life-threatening), or grade 5 (death) adverse event.
Time Frame: From birth through week 26
Population: Live-born infants from PrEP Comparison Component were included in the analysis. Primary analyses, as described in the SAP, were conducted in two groups: PrEP-exposed and PrEP-unexposed. Cohort 1 and Cohort 2/Step 2 were combined as the PrEP-exposed group. The incidence of adverse events was calculated per 100 person-years. Infant participants in Cohort 2/Step 2 contributed to person-years for both groups, with Cohort 2/Step 1 censored upon enrollment in Step 2.
Measure: Number (95% Confidence Interval); unit: number of new cases per 100 person years
Groups:
- Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2): Infants born to women in PrEP Comparison Cohort 1 or Cohort 2/Step 2. Infants did not directly receive PrEP, but may have been exposed to PrEP through placental or breastmilk transfer.
- Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1): Infants born to women in PrEP Comparison Cohort 2/Step 1. Infants were not exposed to PrEP during the study.
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 230 | 112
number of new cases per 100 person years | 42.6 [29.6 to 61.2] | 33.1 [18.4 to 59.7]
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); The incidence rate ratio of cumulative infant AEs between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed (Cohort 2/Step 1) reference group was based on incidence per person-time follow-up. Cohort 2/Step 2 infants contributed person-time to both Cohort 2/Step 1 and Step 2; Test type: Other; Incidence rate ratio = 1.29, 95% CI 2-sided [0.70 to 2.38]

13. Primary Outcome: Mean Infant Bone Mineral Content of Whole Body at Birth
Description: Infant bone mineral content was measured by a dual-energy x-ray absorptiometry (DXA) scan of the whole body (WB-BMC)
Time Frame: Measured at birth
Population: Infants from PrEP Comparison Component with available DXA data were included in this analysis. Primary analyses, as described in the SAP, were conducted in two groups: PrEP-exposed and PrEP-unexposed. Cohort 1 and Cohort 2/Step 2 were combined as the PrEP-exposed group.
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 128 | 74
gram | 68.2 (13.3) | 65.8 (12.0)
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); A two-sample t-test was used to evaluate the difference in mean infant whole-body bone mineral content (WB-BMC) at birth between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed group (Cohort 2/Step 1); Test type: Other; p = 0.18, t-test, 2 sided

14. Primary Outcome: Mean Infant Bone Mineral Content of Lumbar Spine at Birth
Description: Infant bone mineral content was measured by a dual-energy x-ray absorptiometry (DXA) scan of the lumbar spine (LS-BMC)
Time Frame: Measured at birth
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 107 | 73
gram | 1.9 (0.5) | 1.8 (0.4)
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); A two-sample t-test was used to evaluate the difference in mean infant lumbar-spine bone mineral content (WB-BMC) at birth between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed group (Cohort 2/Step 1); Test type: Other; p = 0.39, t-test, 2 sided

15. Primary Outcome: Mean Infant Bone Mineral Content of Lumbar Spine at Week 26
Description: Infant bone mineral content was measured by a dual-energy x-ray absorptiometry (DXA) scan of the lumbar spine (LS-BMC)
Time Frame: Measured at week 26 post-birth
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 131 | 48
gram | 3.2 (0.6) | 3.1 (0.7)
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); A two-sample t-test was used to evaluate the difference in mean infant lumbar-spine bone mineral content (WB-BMC) at week 26 between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed group (Cohort 2/Step 1); Test type: Other; p = 0.12, t-test, 2 sided

16. Primary Outcome: Mean Infant Creatinine Levels at Birth in the PrEP Comparison Component
Description: Infant creatinine levels were obtained from the chemistry/hematology test results at the birth visit
Time Frame: Measured at birth
Population: Infants from PrEP Comparison Component with available creatinine data were included in this analysis. Primary analyses, as described in the SAP, were conducted in two groups: PrEP-exposed and PrEP-unexposed. Cohort 1 and Cohort 2/Step 2 were combined as the PrEP-exposed group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 192 | 95
mg/dL | 0.4 (0.2) | 0.3 (0.1)
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); A two-sample t-test was used to evaluate the difference in mean infant creatinine levels at birth between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed group (Cohort 2/Step 1); Test type: Other; p = 0.70, t-test, 2 sided

17. Primary Outcome: Mean Infant Creatinine Levels at Week 26 in the PrEP Comparison Component
Description: Infant creatinine levels were obtained from the chemistry/hematology test results at week 26 visit
Time Frame: Measured at week 26 post-birth
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 206 | 87
mg/dL | 0.2 (0.0) | 0.2 (0.0)
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); A two-sample t-test was used to evaluate the difference in mean infant creatinine levels at week 26 between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed group (Cohort 2/Step 1); Test type: Other; p = 0.58, t-test, 2 sided

18. Primary Outcome: Mean Infant Creatinine Clearance (CrCl) Rate at Birth in the PrEP Comparison Component
Description: The infant creatinine clearance (CrCl) rate was calculated using creatinine levels and length based on the Schwartz equation.
Time Frame: Measured at birth
Population: Infants from PrEP Comparison Component with available creatinine clearance data were included in this analysis. Primary analyses, as described in the SAP, were conducted in two groups: PrEP-exposed and PrEP-unexposed. Cohort 1 and Cohort 2/Step 2 were combined as the PrEP-exposed group.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 192 | 95
mL/min | 84.4 (61.6) | 74.6 (33.7)
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); A two-sample t-test was used to evaluate the difference in mean infant creatinine clearance rate at birth between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed group (Cohort 2/Step 1); Test type: Other; p = 0.08, t-test, 2 sided

19. Primary Outcome: Mean Infant Creatinine Clearance (CrCl) Rate at Week 26 in the PrEP Comparison Component
Description: as for outcome 18
Time Frame: Measured at week 26 post-birth
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 205 | 86
mL/min | 143.3 (42.5) | 140.1 (37.3)
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); A two-sample t-test was used to evaluate the difference in mean infant creatinine clearance rate at week 26 between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed group (Cohort 2/Step 1); Test type: Other; p = 0.52, t-test, 2 sided

20. Primary Outcome: Mean Infant Length-for-age Z-score at Birth
Description: The infant length-for-age Z-score was calculated based on the infant's sex, length, and age (in days) using WHO child growth standards. The Z-scores range from a minimum of -6 to a maximum of +6. Higher Z-scores indicate better outcomes, reflecting closer adherence to the WHO standards for infant length-for-age. A Z-score of 0 means that the infant's length is exactly at the mean length of the reference population. Z-score between -2 and +2 is considered normal or average. Infants within this range are typically seen as having an appropriate length for their age. Z-score < -3 is a threshold to identify severe stunting, indicating that the infant's length is significantly below the average and pointing to severe chronic undernutrition or other serious health concerns.
Time Frame: Measured at birth
Population: Infants from PrEP Comparison Component with available length-for-age z-score data were included in this analysis. Primary analyses, as described in the SAP, were conducted in two groups: PrEP-exposed and PrEP-unexposed. Cohort 1 and Cohort 2/Step 2 were combined as the PrEP-exposed group.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 197 | 97
Z-score | -0.4 (1.4) | -0.6 (1.2)
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); A two-sample t-test was used to evaluate the difference in mean infant length-for-age z-score at birth between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed group (Cohort 2/Step 1); Test type: Other; p = 0.30, t-test, 2 sided

21. Primary Outcome: Mean Infant Length-for-age Z-score at Week 26
Description: as for outcome 20
Time Frame: Measured at week 26 post-birth
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) | Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1)
Number analyzed (Participants) | 205 | 87
Z-score | -0.6 (1.2) | -0.8 (1.1)
Statistical Analysis 1: Comparison: Infant PrEP Comparison PrEP-Exposed (Cohort 1 and Cohort 2/Step 2) vs Infant PrEP Comparison PrEP-Unexposed (Cohort 2/Step 1); A two-sample t-test was used to evaluate the difference in mean infant length-for-age z-score at week 26 between PrEP-exposed group (Cohort 1 and Cohort 2/Step 2) and PrEP-unexposed group (Cohort 2/Step 1); Test type: Other; p = 0.06, t-test, 2 sided

22. Secondary Outcome: Maternal Median Steady State TFV-DP Concentration Levels at Study Week 12 During Pregnancy and Postpartum
Description: TFV-DP concentration levels were measured using dried blood spots (DBS). Concentrations measured at week 12 represent the steady-state TFV-DP concentration.
Time Frame: Assessed at study Week 12 during pregnancy for Maternal PK Component Group 1 and at study Week 12 during postpartum for Maternal PK Component Group 2
Population: Evaluable participants from PK Components were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: fmol/punch
Arm/Group | Maternal PK Component Group 1 | Maternal PK Component Group 2
Number analyzed (Participants) | 20 | 20
fmol/punch | 965 [691 to 1166] | 1406 [1053 to 1859]
Statistical Analysis 1: Comparison: Maternal PK Component Group 1 vs Maternal PK Component Group 2; Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: For women, adverse events were reported from enrollment to the end of study follow-up (26 weeks postpartum), up to one year. For infants, adverse events were reported from birth to the end of study follow-up (26 weeks after birth).
Description: Grade 3 or higher, serious, and targeted lower grade adverse events (AEs) were reported for all enrolled women and live-born infants using the DAIDS AE Grading Table (July 2017).
Arm/Group | Maternal PK Component Group 1 | Maternal PK Component Group 2 | Maternal PrEP Comparison Cohort 1 | Maternal PrEP Comparison Cohort 2/Step 1 | Maternal PrEP Comparison Cohort 2/Step 2 | Infant PK Component Group 1 | Infant PK Component Group 2 | Infant PrEP Comparison Cohort 1 | Infant PrEP Comparison Cohort 2/Step 1 | Infant PrEP Comparison Cohort 2/Step 2
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 1/229 | 0/121 | 0/13 | 0/18 | 0/20 | 9/217 | 5/112 | 0/13
Serious Adverse Events (participants affected / at risk) | 3/20 | 0/20 | 30/229 | 4/121 | 0/13 | 1/18 | 0/20 | 26/217 | 8/112 | 0/13
Other Adverse Events (participants affected / at risk) | 1/20 | 2/20 | 123/229 | 46/121 | 5/13 | 1/18 | 4/20 | 120/217 | 44/112 | 4/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maternal PK Component Group 1 (N=20) | Maternal PK Component Group 2 (N=20) | Maternal PrEP Comparison Cohort 1 (N=229) | Maternal PrEP Comparison Cohort 2/Step 1 (N=121) | Maternal PrEP Comparison Cohort 2/Step 2 (N=13) | Infant PK Component Group 1 (N=18) | Infant PK Component Group 2 (N=20) | Infant PrEP Comparison Cohort 1 (N=217) | Infant PrEP Comparison Cohort 2/Step 1 (N=112) | Infant PrEP Comparison Cohort 2/Step 2 (N=13)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Birth mark (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroschisis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperprolactinaemia (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death neonatal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fever neonatal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 3 | 0
Typhoid fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Apgar score low (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Progesterone decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxic ischaemic encephalopathy neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maternal PK Component Group 1 (N=20) | Maternal PK Component Group 2 (N=20) | Maternal PrEP Comparison Cohort 1 (N=229) | Maternal PrEP Comparison Cohort 2/Step 1 (N=121) | Maternal PrEP Comparison Cohort 2/Step 2 (N=13) | Infant PK Component Group 1 (N=18) | Infant PK Component Group 2 (N=20) | Infant PrEP Comparison Cohort 1 (N=217) | Infant PrEP Comparison Cohort 2/Step 1 (N=112) | Infant PrEP Comparison Cohort 2/Step 2 (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperprolactinaemia (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infantile diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Abscess of external ear (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 7 | 3 | 0 | 0 | 0 | 10 | 2 | 0
Genital ulcer syndrome (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecological chlamydia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mastitis postpartum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 7 | 4 | 0
Ophthalmia neonatorum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Primary syphilis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Puerperal infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 20 | 6 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Septic rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea manuum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Typhoid fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 14 | 6 | 0 | 0 | 0 | 25 | 9 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 21 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginitis chlamydial (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 9 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis chlamydial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Perineal injury (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine cervical laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 10 | 5 | 1
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine renal clearance (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 2 | 17 | 9 | 3 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treponema test positive (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 60 | 15 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Afterbirth pain (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 8 | 2 | 0 | 0 | 0 | 0 | 0 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxic ischaemic encephalopathy neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nipple disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 7 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Neonatal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient neonatal pustular melanosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Episiotomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Therapeutic procedure (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT03386578/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03386578/SAP_001.pdf